CLINICAL TRIAL: NCT03097497
Title: The Effectiveness of a Physiotherapeutic Re-education Based on the Pre-activation of the Transverse Abdominis in Patients With Non-specific Chronic Low Back Pain in Primary Care.
Brief Title: Physiotherapy Re-education of Pre-activation of the Transverse Abdominis in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Francesc Josep Rubi Carnacea, Physiotherapist, Universitat de Lleida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P14/089
Record Dates: First submitted 2017-03-18; First posted 2017-03-31 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Chronic Non-specific Low-Back Pain
Keywords: Chronic Non-specific Low-Back Pain; Chronic Low-Back Pain; Physiotherapy; Therapeutic Exercise; Primary Care; Transverse Abdominal Muscle

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy re-education program (Experimental): Physiotherapy re-education program based on the pre-activation of the transverse abdominal muscle, performed with progressive difficulty and supervised at all times by an expert physiotherapist. The intervention will last 4 weeks, with two weekly sessions of 30-35 minutes each. Sessions will be held individually.
  Interventions: Other: Physiotherapy re-education program
- Conventional treatment by GP (Active Comparator): Will follow conventional treatment prescribed by the general practitioner in a primary care consultation. This conventional treatment is based on the clinical guidlines of the "Institut Català de la Salut"
  http://www.gencat.cat/ics/professionals/guies/docs/guia_lumbalgies.pdf
  Interventions: Other: Conventional treatment by GP

INTERVENTIONS:
Other: Physiotherapy re-education program — Physiotherapy Program based on the Re-education of Pre-activation of the Transverse Abdominal Muscle
  Arms: Physiotherapy re-education program
Other: Conventional treatment by GP — Patients will follow the general practitioner's advice including medication if needed
  Arms: Conventional treatment by GP

SUMMARY:
Hypothesis: The hypothesis of the study is that the physiotherapeutic re-education of the pre-activation of the transverse abdominal muscle decreases pain intensity in patients with chronic non-specific low-back pain by at least 30% and is more effective than conventional treatment.

Aims: the principal aim is to determine the effectiveness of a physiotherapeutic re-education program based on the pre-activation of the transverse abdominal muscle on pain intensity in adult patients diagnosed with chronic non-specific low-back pain compared to conventional treatment in a primary care setting. The secondary aims of the study are to assess the effects of a physiotherapeutic re-education program based on the pre-activation of the transverse abdominal muscle on: (1) disability and limitations for the development of the activities of daily living associated with LBP, (2) transverse abdominal muscle muscle contraction, (3) to assess whether the resistance training parameters applied to older adults are valid for young adults and (4) to determine whether the training protocols used for the cervical spine could be extrapolated to the lumbar spine.

DETAILED DESCRIPTION:
This study will be a parallel randomized controlled trial. Participants between 18-65 years old, diagnosed with chronic nonspecific low-back pain, who will sign the informed consent, will be included in the study. Participants will be excluded if they are diagnosed with cognitive impairments, if the presence of any "Red Flag" is identified, women on pregnancy or postpartum less than three months and participants with difficulties understanding and/or speaking Spanish or Catalan.

Based upon the results of a systematic review about the effectiveness of physical therapy based treatment for low back pain, a reduction in 15 points of pain intensity assessed through Visual Analogue Scale will be considered for sample size calculation. Therefore, accepting an alfa risk of 0.05, a beta risk less than 0.2 and assuming a 15% of withdrawals a sample size of 108 participants has been estimated for this study.

Participants will be recruited from Primary Care Centers of the city of Lleida (Catalonia, Spain). They will be first contacted by telephone and the suitability of each participant will be assessed trough a brief interview. After participant selection via telephone, those who meet the inclusion criteria will be invited to have a personal interview with the researchers in order to solve any doubt and to read and sign the written informed consent. To ensure all participants understand the study, they will simply be asked about general study information (i.e. objectives, treatment and control conditions, etc.).

The included participants will be assigned either to the experimental or the control group using a simple randomization method. The allocation will be concealed to both, the physiotherapists who will make the assessments (pre- and post-treatment and follows-up) of the participants and the researcher who will manage the results data.

Participants in the experimental group will receive an individualized physiotherapeutic re-education program based on the pre-activation of the transverse abdominal muscle. The intervention will last 4-weeks and will consist on two weekly sessions of 30-35 minutes each. Each session will be divided into two main parts (1) warm-up and (2) re-education of the pre-activation of the transverse abdominal muscle.

1. . Warm-up (5 minutes): lumbopelvic dissociation exercises, increasing difficulty each week.
2. . Re-education of the pre-activation of the transverse abdominal muscle (25-30 minutes) First session: participants will learn how to contract appropriately the transverse abdominal muscle through basic and easy exercises. In order to facilitate the contraction, one physiotherapist will monitor the lumbopelvic motion by placing a Pressure Biofeedback Unit under the participants' lumbar spine.

The authors will calculate the 75% of one-rep max (1RM) and the seconds that each participant can maintain the 75% 1RM contraction. This will allow to establish individualized times for carrying out the exercises during the following sessions.

Following sessions: 16 re-educational exercises have been design. In each session, the participants will perform four different exercises, increasing each week the difficulty and the degree of loading. The participants will perform the exercises based on their 75% 1RM calculation, completing 3 series of 9 repetitions, holding each repetition a maximum of 6 seconds. It will be a pause of 4 sec. between each exercise and a pause of 60 seconds between each series. The 75% 1RM will be calculated in each session.

Participants in the control group will follow the conventional treatment prescribe by their general practitioner in primary care.

Participants in both groups will be assessed pre- and post-treatment with a follow-up at 3, 6 and 12 months.

All statistical analyses will be carried out using the statistical program 'PASW 20'. An intention to treat analysis will be performed.

Expected outcomes: the authors expect that patients in the experimental group will achieve a greater (1) reduction in pain intensity, (2) improvement of disability associated with CLBP, (3) improvement in the development of activities of daily living, and (4) contraction of the transvers abdominal muscle, compared to patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed of non-specific chronic low back pain of 3 or more months duration.
2. Patients between 18-65 years old.
3. To accept and sign the informed consent.

Exclusion Criteria:

1. Patients with diagnosed of cognitive problems that prevent understanding the procedure or participation in the study.
2. Any red flag condition:

   * Age of pain onset <20 or >55
   * Recent history of trauma
   * Pain not associated with movement and not relieved by lying down
   * Thoracic pain
   * Past history of malignancy, recurrent of prolonged use of corticosteroids, immunosuppression/HIV
   * Being systematically unwell
   * Unexplained weight loss
   * Neurological symptoms such as weakness of the limbs
   * Structural deformity of the spine
3. Women on pregnancy or postpartum less than three months.
4. Difficulty understanding and/or speaking Spanish or Catalan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity (from baseline) | 4 weeks, 3 months, 6 months, 12 months
  The Visual Analogue Scale (VAS) is an unidimensional scale developed to measure pain intensity. This scale consists on a line of 100-mm with a description on both extremes. "No pain" appears on the left side, representing a value of 0, and "worst pain ever" appears on the right side of the scale, representing a value of 100. A higher score on the scale will be indicative of greater pain intensity. Although no normative values are available in regard of the distribution of VAS scores, the following cut-off scores have been recommended: no pain (0-4mm), slight pain (5-44mm), moderate pain (45-74mm) and severe pain (75-100mm)

SECONDARY OUTCOMES:
Oswestry Disability Index | 4 weeks, 3 months, 6 months, 12 months
  The Oswestry Disability Index (ODI) was created by John O'Brien (1976). It is a self-administered questionnaire that allows assessing the degree of disability and the limitations in activities of daily living related to low back pain.
  The ODI contains ten main topics regarding pain intensity, lifting, self-care ability, sleep quality, social life, ability to sit, stand and walk, ability to travel and sexual function. This index consists of 10 questions with six potential responses scored from 0 to 5.
  The measurement percentages are:
  * 0-19%: minimal disability
  * 20-39%: moderate disability
  * 40-59%: intense disability
  * 60-79%: severe disability
  * 80-100%: maximal disability
Roland-Morris Scale | 4 weeks, 3 months, 6 months, 12 months
  The Roland-Morris Scale (RMS) determines the degree of physical disability derived from nonspecific low back pain. It especially detects cases in which the degree of disability is exaggeratedly high or persistent. In order to establish the degree of disability, the numbers of items selected by each patient are counted, with the score ranging from 0 (absence of disability) to 24 (maximum degree of disability). A total score below 4 points is categorized as mild impairment. In monitoring patients' progress, a change of 2 points or more is considered as relevant.
Transverse abdominal muscle contraction with Pressure Biofeedback Unit | 4 weeks, 3 months, 6 months, 12 months
  The Pressure Biofeedback Unit (PBU) is a simple pressure transducer consisting of a pressure cushion with three air filled chambers and connected to a sphygmomanometer. The pressure bag is 17.7 x 24 cm size and is made of inelastic material. The scale measured with the sphygmomanometer goes from 0mmHg to 200mmHg. The PBU registers the pressure caused by movement or change of position and is used to obtain information on the effect of a muscle contraction. Research on PBU indicates that it is a valid tool for measuring transverse abdominal muscle activity in people with non-specific chronic low back pain and has an intra- and inter-examiner agreement of a 95%.
Surface Electromyography | 4 weeks, 3 months, 6 months, 12 months
  Surface electromyography is a method of recording the electrical-physiological activity generated after a muscle contraction. It is, therefore, a method of quantitative and non-invasive assessment that allows capturing the action potentials produced by the muscles of the explored zone. The electrical signal is captured by one or more electrodes placed strategically on the surface of the skin and sent to a receiving device for its processing. Thus, obtaining a frequency and intensity that allow us to interpret what is happening at the muscular level in different situations.
  The electrodes used have a diameter of 10mm and should be placed in the cutaneous zone adjacent to the assessed musculature. Frequencies range from 20 to 500 Hz.
  The most important parameters that can be extracted are timing and intensity of muscle activation as well as muscle fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Francesc J Rubí Carnacea, PhDc, Principal Investigator — Universitat de Lleida; Jorge Soler González, GP, Study Director — Universitat de Lleida
Locations (1):
- Primary care setting, Lleida, Spain

REFERENCES:
- [Derived] Rubi-Carnacea F, Masbernat-Almenara M, Climent-Sanz C, Soler-Gonzalez J, Garcia-Escudero M, Martinez-Navarro O, Valenzuela-Pascual F. Effectiveness of an exercise intervention based on preactivation of the abdominal transverse muscle in patients with chronic nonspecific low back pain in primary care: a randomized control trial. BMC Prim Care. 2023 Sep 6;24(1):180. doi: 10.1186/s12875-023-02140-3. PMID 37674205